CLINICAL TRIAL: NCT05838313
Title: Should I Have an Elective Induction? The SELECTION Study
Brief Title: Should I Have an Elective Induction?
Acronym: SELECTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Ohio State University (Other); University of California, San Francisco (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY004944; R21HD098496 (NIH)
Record Dates: First submitted 2022-12-13; First posted 2023-05-01 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Labor, Induced; Patient Preference
Keywords: Shared Decision Making
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision Support Tool (Experimental): Participants will interact with the decision support tool prior to making their decision regarding whether to have an induction of labor without a medical indication
  Interventions: Behavioral: Elective Induction of Labor Decision Support Tool

INTERVENTIONS:
Behavioral: Elective Induction of Labor Decision Support Tool — Decision support tool for people having their first baby and planning vaginal delivery without a medical indication for induction of labor

SUMMARY:
The goal of the proposed study is to perform a pilot test of a patient-centered decision support tool to help pregnant people and providers work together in making informed, shared decisions regarding whether or not to opt for elective IOL at 39 weeks gestation

DETAILED DESCRIPTION:
60 nulliparous pregnant people with singleton, vertex pregnancies at 36-38 weeks who do not have an indication for induction of labor (IOL) will be enrolled and will view a decision support tool (DST) regarding induction without medical indication. During the enrollment face-to-face interview, participants will interact with the DST and complete pre- and post-DST viewing questionnaires. The investigators will conduct telephone interviews a few days later but before 39+0 weeks, and again 2-4 weeks postpartum and will review the medical record for delivery events and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant person
* Nulliparous
* Planned vaginal delivery
* No medical indication for induction of labor

Exclusion Criteria:

* Contraindication to vaginal delivery
* Prior delivery (vaginal or cesarean)
* Medical indication for induction of labor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of South Florida, Tampa, Florida
  - The Ohio State University, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Decision Support Tool
Started | 66
Completed | 66
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 39
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 66

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: Recruitment rate, defined as the number of people who agree to participate out of those who are approached for the study
Time Frame: 32-38 weeks gestation
Population: Recruitment rate will be calculated based on the number of people approached who were eligible and agreed to participate in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 176
Participants | 66

2. Primary Outcome: Proportion of People Completely Viewing the Decision Support Tool
Description: The proportion of participants who view all of the pages of the decision support tool will be calculated
Time Frame: 36-38 weeks gestation
Population: All participants interacting with the decision support tool
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 66
Participants | 52

3. Secondary Outcome: Satisfaction With the Decision Support Tool
Description: 4 item scale. Range of 0-20, with higher scores indicating higher satisfaction.
Time Frame: 36-38 weeks gestation
Population: Participants completing questionnaire after interacting with the decision support tool
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 66
score on a scale | 17.4 (2.7)

4. Secondary Outcome: Satisfaction With the Decision Support Tool
Description: 4 item scale. Range of 0-20, with higher scores indicating higher satisfaction.
Time Frame: 38-39 weeks gestation, prior to delivery
Population: Participants completing follow up questionnaire at 38-39 weeks gestation, prior to delivery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 49
score on a scale | 17.0 (3.0)

5. Secondary Outcome: Impact of App on Decision Making
Description: 5 point scale (Strongly disagree to Strongly agree, 5=Strongly agree) "Viewing the App affected my decision making"
Time Frame: 2-4 weeks Postpartum
Population: Participants completing follow up questionnaire at 2-4 weeks postpartum
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 52
units on a scale | 2.8 (1.1)

ADVERSE EVENTS:
Time Frame: From study start through completion of the last chart review (30 weeks)
Arm/Group | Decision Support Tool
All-Cause Mortality (participants affected / at risk) | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66
Other Adverse Events (participants affected / at risk) | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT05838313/Prot_SAP_000.pdf